CLINICAL TRIAL: NCT04271098
Title: Risk Factors, Hepatic Dysfunction, and Open-heart Surgery
Brief Title: The Investigation of the Causes of Hepatic Dysfunction in the Postoperative Period During Open-heart Surgeries
Status: Completed | Type: Observational
Sponsor: Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ayse Baysal, Associate Professor, Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital
Other Study IDs: 2011.3/05
Record Dates: First submitted 2020-02-11; First posted 2020-02-17 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Hyperbilirubinemia; Hepatic Impairment; Surgery; Cardiac Disease
Keywords: open-heart surgery; postoperative; complications; hyperbilirubinemia; hepatic impairment
MeSH Terms: conditions — Hyperbilirubinemia; Heart Diseases | interventions — Time

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Open-heart surgery: Patients undergoing open-heart surgery with cardiopulmonary bypass
  Interventions: Procedure: Open-Heart Surgery for nine months duration; Other: Relation between possible risk factors and hyperbilirubinemia; Other: Follow-up period

INTERVENTIONS:
Procedure: Open-Heart Surgery for nine months duration — In a single group of patients including 340 patients undergoing open-heart surgery during a period of nine months, the collected parameters include; alanine transaminase (ALT), aspartate transaminase (AST), alkaline phosphatase (ALP), total bilirubin (TBIL), and gamma-glutamyl transpeptidase (GGT) and albumin preoperatively and on postoperative days of 1, 3 and 7. All patients were divided into two groups as with or without hyperbilirubinemia, and this was defined by the occurrence of a plasma total bilirubin concentration of more than 34 µmol/L (2 mg/dL) in any measurement during the postoperative period. For each diagnostic test, a comparison within the group for different time points was statistically evaluated by analysis of variance tests.
  Other Names: Type of open-heart surgical operation (coronary artery bypass graft operation, mitral valve, aortic valve or multiple valvular surgeries); Hyperbilirubinemia; Hepatic function related tests
Other: Relation between possible risk factors and hyperbilirubinemia — Possible preoperative, intraoperative, and postoperative risk factors were investigated. The relations between hyperbilirubinemia and possible risk factors are sought by the use of the statistical analysis methods including logistic regression analysis.
Other: Follow-up period — All patients were investigated for a period of ten days postoperatively. During this period, intensive care unit (ICU) stay, in-hospital stay, and all adverse events were recorded.

SUMMARY:
In a prospective observational study during the six-month duration, coronary artery bypass graft surgery (CABG) and valve repair surgery (mitral, mitral, and aortic valve and/or tricuspid valve) patients were investigated for hepatic dysfunction. All patients were divided into two groups as with or without hyperbilirubinemia, and this was defined by the occurrence of a plasma total bilirubin concentration of more than 34 µmol/L (2 mg/dL) in any measurement during the postoperative period. Our goal was to determine the risk factors associated with hepatic dysfunction in patients undergoing open-heart surgery with cardiopulmonary bypass. The collected parameters include; alanine transaminase (ALT), aspartate transaminase (AST), alkaline phosphatase (ALP), total bilirubin (TBIL), and gamma-glutamyl transpeptidase (GGT) and albumin preoperatively and on postoperative days 1, 3 and 7. Possible preoperative, intraoperative, and postoperative risk factors were investigated. Logistic regression analysis was done to identify the risk factors for postoperative hyperbilirubinemia.

DETAILED DESCRIPTION:
There are a series of pathophysiological changes in patients undergoing open-heart surgeries with cardiopulmonary bypass (CPB) that causes liver hypoperfusion, centrilobular sinusoid ischemia, and subsequent reperfusion injuries, hemolysis, or systemic inflammatory response. These events may eventually lead to various forms of hepatic dysfunction in patients during the postoperative period after open-heart surgeries. An increased incidence of liver function test abnormalities were reported, and the rates vary between 10 % and 40%. The occurrence of postoperative hyperbilirubinemia is crucial in increased morbidity and mortality after open-heart surgery with CPB. There are several reports of the possible risk factors that are associated with hepatic dysfunction. In previous studies, the incidence of postoperative hyperbilirubinemia was between the range of 20% up to 51% in open-heart surgeries with CPB. The causes of this higher incidence were related to the presence of various possible risk factors, and these include; valvular heart disease and related low cardiac output states, and low ejection fraction. Other important risk factors for postoperative hepatic dysfunction after open-heart surgery with CPB were longer operative time and a larger volume of blood transfusion. However, CPB itself is not a significant constituent in the postoperative development of hyperbilirubinemia. Splanchnic ischemia before or during operation and in the postoperative period appears to be an essential cause. Other risk factors that were identified as possible risk factors for postoperative hepatic dysfunction. We can list these factors as; poor preoperative heart function, hemodynamic instability, emergency surgery, and preoperative liver dysfunction. Our goal was to determine the possible risk factors associated with hepatic dysfunction in patients undergoing open-heart surgery with CPB.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing open-heart surgery with CPB,
* Patients between the ages of 19 to 80,
* American Society of Anesthesiologist (ASA) status of 2 and 3,
* Preoperative ejection fraction (EF) greater than 30%.
* There were five different open-heart surgery group of patients in this study. The groups include; coronary artery bypass grafting (CABG), mitral valvular replacement, aortic valvular replacement, combined mitral and aortic valve replacement, combined mitral, aortic and/or tricuspid valve replacements.

Exclusion Criteria:

* Both CABG and valve replacement,
* Resection of a ventricular or aortic aneurysm,
* Transplantation or another surgical procedure,
* Reoperation of valvular repair surgery, patients with preoperative ejection fraction less than 30%,
* Preoperative hyperbilirubinemia defined as total bilirubin concentration of more than 3 mg/dL,
* Preoperative congestive heart failure, preoperative renal dysfunction (serum creatinine greater than 1.3 mg/dL),
* Chronic oliguria/anuria requiring dialysis,
* Preoperative American Society of Anesthesiologist (ASA) status of 4,
* History of pancreatitis or current corticosteroid treatment.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is performed on a patient population undergoing open-heart surgery with cardiopulmonary bypass.
Sampling Method: Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2012-07-01 (Actual); Study Completion 2012-09-01 (Actual)

PRIMARY OUTCOMES:
Comparison of serum total bilirubin values on postoperative day 1. | Preoperative one day before surgery and postoperative day 1.
  Change from baseline (preoperative) of serum total bilirubin on postoperative day 1.
Comparison of serum total bilirubin values on postoperative day 3. | Preoperative one day before surgery and postoperative day 3.
  Change from baseline (preoperative) of serum total bilirubin on postoperative day 3.
Comparison of serum total bilirubin values on postoperative day 7. | Preoperative one day before surgery and postoperative day 7.
  Change from baseline (preoperative) of serum total bilirubin on postoperative day 7.
Comparison of all serum total bilirubin values at all collected times. | Preoperatively one day before surgery and on postoperative days of 1, 3 and 7.
  A repeated measures statistical analysis using analysis of variance tests was performed.
Comparison of serum albumin values on postoperative day 1. | Preoperative one day before surgery and postoperative day 1.
  Change from baseline (preoperative) of serum albumin on postoperative day 1.
Comparison of serum albumin values on postoperative day 3. | Preoperative one day before surgery and postoperative day 3.
  Change from baseline (preoperative) of serum albumin on postoperative day 3.
Comparison of serum albumin values on postoperative day 7. | Preoperative one day before surgery and postoperative day 7.
  Change from baseline (preoperative) of serum albumin on postoperative day 7.
Comparison of all serum albumin values at all collected times. | Preoperatively one day before surgery and on postoperative days of 1, 3 and 7.
  A repeated measures statistical analysis using analysis of variance tests was performed.
Comparison of serum alkaline phosphatase (ALP) values on postoperative day 1. | Preoperative one day before surgery and on postoperative day of 1.
  Change from baseline (preoperative) of serum alkaline phosphatase (ALP) on postoperative day 1.
Comparison of serum alkaline phosphatase (ALP) values on postoperative day 3. | Preoperative one day before surgery and on postoperative day of 3.
  Change from baseline (preoperative) of serum alkaline phosphatase (ALP) on postoperative day 3.
Comparison of serum alkaline phosphatase (ALP) values on postoperative day 7. | Preoperative one day before surgery and on postoperative day of 7.
  Change from baseline (preoperative) of serum alkaline phosphatase (ALP) on postoperative day 7.
Comparison of all serum alkaline phosphatase (ALP) values at all collected times. | Preoperatively one day before surgery and on postoperative days of 1, 3 and 7.
  A repeated measures statistical analysis using analysis of variance tests was performed.
Comparison of serum alanine transaminase (ALT) values on postoperative day 1. | Preoperatively one day before surgery and on postoperative day of 1.
  Change from baseline (preoperative) of serum alanine transaminase (ALT) on postoperative day 1.
Comparison of serum alanine transaminase (ALT) values on postoperative day 3. | Preoperatively one day before surgery and on postoperative day of 3.
  Change from baseline (preoperative) of serum alanine transaminase (ALT) on postoperative day 3.
Comparison of serum alanine transaminase (ALT) values on postoperative day 7. | Preoperatively one day before surgery and on postoperative day of 7.
  Change from baseline (preoperative) of serum alanine transaminase (ALT) on postoperative day 7.
Comparison of all serum alanine transaminase (ALT) values at all collected times. | Preoperatively one day before surgery and on postoperative days of 1, 3 and 7.
  A repeated measures statistical analysis using analysis of variance tests was performed.
Comparison of serum aspartate transaminase (AST) values on postoperative day 1. | Preoperatively one day before surgery and on postoperative day of 1.
  Change from baseline (preoperative) of serum aspartate transaminase (AST) on postoperative day 1.
Comparison of serum aspartate transaminase (AST) values on postoperative day 3. | Preoperatively one day before surgery and on postoperative day of 3.
  Serum aspartate transaminase (AST) values were collected preoperative and postoperative day 3.
Comparison of serum aspartate transaminase (AST)values on postoperative day 7. | Preoperatively one day before surgery and on postoperative day of 7.
  Serum aspartate transaminase (AST) values were collected preoperative and postoperative day 7.
Comparison of all serum aspartate transaminase (AST) values at all collected times. | Preoperatively one day before surgery and on postoperative days of 1, 3 and 7.
  A repeated measures statistical analysis using analysis of variance tests was performed.
Comparison of serum lactate dehydrogenase (LDH) values on postoperative day 1. | Preoperatively one day before surgery and on postoperative day of 1.
  Change from baseline (preoperative) of serum lactate dehydrogenase (LDH) on postoperative day 1.
Comparison of serum lactate dehydrogenase (LDH) values on postoperative day 3. | Preoperatively one day before surgery and on postoperative day of 3.
  Change from baseline (preoperative) of serum lactate dehydrogenase (LDH) on postoperative day 3.
Comparison of serum lactate dehydrogenase (LDH) values on postoperative day 7. | Preoperatively one day before surgery and on postoperative day of 7.
  Change from baseline (preoperative) of serum lactate dehydrogenase (LDH) on postoperative day 7.
Comparison of all serum lactate dehydrogenase (LDH) values at collected times. | Preoperatively one day before surgery and on postoperative days of 1, 3 and 7.
  A repeated measures statistical analysis using analysis of variance tests was performed.
Comparison of serum glutamyl transpeptidase (GGT) values on postoperative day 1. | Preoperatively one day before surgery and on postoperative day of 1.
  Change from baseline (preoperative) of serum glutamyl transpeptidase (GGT) on postoperative day 1.
Comparison of serum glutamyl transpeptidase (GGT) values on postoperative day 3. | Preoperatively one day before surgery and on postoperative day of 3.
  Change from baseline (preoperative) of serum glutamyl transpeptidase (GGT) on postoperative day 3.
Comparison of serum glutamyl transpeptidase (GGT) values on postoperative day 7. | Preoperatively one day before surgery and on postoperative day of 7.
  Change from baseline (preoperative) of serum glutamyl transpeptidase (GGT) on postoperative day 7.
Comparison of all serum glutamyl transpeptidase (GGT) values at collected times. | Preoperatively one day before surgery and on postoperative days of 1, 3 and 7.
  A repeated measures statistical analysis using analysis of variance tests was performed.

SECONDARY OUTCOMES:
Use of aortic cross-clamp time; as a risk factor | During intraoperative time
  Use of aortic cross-clamp time
Use of cardiopulmonary bypass time; as a risk factor | During intraoperative time
  Use of cardiopulmonary bypass time
Use of inotropic support; as a risk factor | During intraoperative time and in the first 10 days of postoperative period
  Use of various inotropic support agents
Use of intra-aortic balloon pump; as a risk factor | During intraoperative time and in the first 10 days of postoperative period
  Use of intra-aortic balloon pump
Use of prolonged mechanical ventilation; as a risk factor | During the first 30 days of postoperative period
  Duration of prolonged mechanical ventilation
Development of pneumonia; as a risk factor | During the first 10 days of postoperative period
  Presence of development of pneumonia
Development of perioperative heart attack; a rsik factor | During intraoperative time and in the first 10 days of postoperative period
  Presence of perioperative myocardial infarction
Cerebrovascular event; a risk factor | During the first 10 days of postoperative period
  Development of cerebrovascular event (stroke, transient ischemic attack), seizure
Presence of rhythm disturbance; a risk factor | During intraoperative time and in the first 10 days of postoperative period
  Presence of atrial fibrillation and other rhythm disturbances
Need of renal replacement therapy; a risk factor | During the first 10 days of postoperative period
  Need for renal replacement therapy (RRT)
Need of reoperation; a risk factor | During the first 10 days of postoperative period
  Need of reoperation secondary to bleeding
Presence of other adverse events; a risk factor | During the first 10 days of postoperative period
  Presence of other adverse events such as; development of sepsis or need for tracheostomy
Duration of intensive care unit stay; a risk factor | During the first 10 days of postoperative period
  Duration of intensive care unit stay
Duration of in-hospital stay; a risk factor | During the first 30 days of postoperative period
  Duration of in-hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Baysal, MD, Principal Investigator — Pendik Bolge Hospital

IPD SHARING:
Plan to Share IPD: Yes
We can share the study protocol, clinical study report, the excel data of our clinical work.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data is available upon registration and it will be available on the web site if needed.
Access Criteria: Accessible to all researchers.

REFERENCES:
- [Background] Zhou W, Wang G, Liu Y, Tao Y, Du Z, Tang Y, Qiao F, Liu Y, Xu Z. Outcomes and risk factors of postoperative hepatic dysfunction in patients undergoing acute type A aortic dissection surgery. J Thorac Dis. 2019 Aug;11(8):3225-3233. doi: 10.21037/jtd.2019.08.72. PMID 31559024
- [Result] Wang MJ, Chao A, Huang CH, Tsai CH, Lin FY, Wang SS, Liu CC, Chu SH. Hyperbilirubinemia after cardiac operation. Incidence, risk factors, and clinical significance. J Thorac Cardiovasc Surg. 1994 Sep;108(3):429-36. PMID 8078336
- [Result] Michalopoulos A, Alivizatos P, Geroulanos S. Hepatic dysfunction following cardiac surgery: determinants and consequences. Hepatogastroenterology. 1997 May-Jun;44(15):779-83. PMID 9222689
- [Result] Lockey E, McIntyre N, Ross DN, Brookes E, Sturridge MF. Early jaundice after open-heart surgery. Thorax. 1967 Mar;22(2):165-9. doi: 10.1136/thx.22.2.165. PMID 6033384
- [Result] Collins JD, Bassendine MF, Ferner R, Blesovsky A, Murray A, Pearson DT, James OF. Incidence and prognostic importance of jaundice after cardiopulmonary bypass surgery. Lancet. 1983 May 21;1(8334):1119-23. doi: 10.1016/s0140-6736(83)92863-5. PMID 6133152
- [Result] Chu CM, Chang CH, Liaw YF, Hsieh MJ. Jaundice after open heart surgery: a prospective study. Thorax. 1984 Jan;39(1):52-6. doi: 10.1136/thx.39.1.52. PMID 6695353
- [Result] Naschitz JE, Slobodin G, Lewis RJ, Zuckerman E, Yeshurun D. Heart diseases affecting the liver and liver diseases affecting the heart. Am Heart J. 2000 Jul;140(1):111-20. doi: 10.1067/mhj.2000.107177. PMID 10874271
- [Result] McSweeney ME, Garwood S, Levin J, Marino MR, Wang SX, Kardatzke D, Mangano DT, Wolman RL; Investigators of the Ischemia Research and Education Foundation and the Multicenter Study of Perioperative Ischemia Research Group. Adverse gastrointestinal complications after cardiopulmonary bypass: can outcome be predicted from preoperative risk factors? Anesth Analg. 2004 Jun;98(6):1610-1617. doi: 10.1213/01.ANE.0000113556.40345.2E. PMID 15155313
- [Result] D'Ancona G, Baillot R, Poirier B, Dagenais F, de Ibarra JI, Bauset R, Mathieu P, Doyle D. Determinants of gastrointestinal complications in cardiac surgery. Tex Heart Inst J. 2003;30(4):280-5. PMID 14677737
- [Result] Atoui R, Ma F, Langlois Y, Morin JF. Risk factors for prolonged stay in the intensive care unit and on the ward after cardiac surgery. J Card Surg. 2008 Mar-Apr;23(2):99-106. doi: 10.1111/j.1540-8191.2007.00564.x. PMID 18304122
- [Result] Sharma P, Ananthanarayanan C, Vaidhya N, Malhotra A, Shah K, Sharma R. Hyperbilirubinemia after cardiac surgery: An observational study. Asian Cardiovasc Thorac Ann. 2015 Nov;23(9):1039-43. doi: 10.1177/0218492315607149. Epub 2015 Sep 23. PMID 26405017